CLINICAL TRIAL: NCT02382497
Title: New Treatment Perspectives in Eating Disorders: the Efficacy of Non-invasive Brain-directed Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mariella Enoc (Other)
Responsible Party: Sponsor-Investigator, Mariella Enoc, Responsible of the Child Neuropsychiatry Unit, Bambino Gesù Hospital and Research Institute
Organization: Bambino Gesù Hospital and Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 763_OPBG_2014
Record Dates: First submitted 2015-02-27; First posted 2015-03-06 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Eating Disorders; Binge Eating Disorder; Anorexia Nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Binge-Eating Disorder; Anorexia Nervosa

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AN Active tDCS (Experimental): Treatment "as usual" plus experimental treatment
  Interventions: Device: AN Active tDCS
- AN Sham tDCS (Sham Comparator): Treatment "as usual" plus placebo treatment
  Interventions: Device: AN Sham tDCS
- BED Active tDCS (Experimental): Treatment "as usual" plus experimental treatment
  Interventions: Device: BED Active tDCS
- BED Sham tDCS (Sham Comparator): Treatment "as usual" plus placebo treatment
  Interventions: Device: BED Sham tDCS

INTERVENTIONS:
Device: AN Active tDCS — The tDCS active stimulations will be directed to PFC regions for six weeks delivered for three times a week.
  tDCS will be delivered by a battery driven, constant current stimulator through a pair of saline-soaked sponge electrodes kept firm by elastic bands.
  The anode will be placed on the left PFC, F3 position according to the 10-20 international EEG system for electrode placement, while the cathode will be placed on the right PFC, F4 position according to the 10-20 international EEG system for electrode placement.
  Stimulation intensity will be set at 1 milliampere (mA), the duration of stimulation will be 20 min.
  Other Names: Brain Stim
  Arms: AN Active tDCS
Device: AN Sham tDCS — The same electrode placement will be used as in the stimulation conditions (left anodal/right cathodal), but the current will be applied for 30 s and will be ramped down without the participants awareness, and will be held three times a week for six weeks.
  Other Names: Brain Stim Sham
  Arms: AN Sham tDCS
Device: BED Active tDCS — The tDCS active stimulations will be directed to PFC regions for six weeks delivered for three times a week.
  tDCS will be delivered by a battery driven, constant current stimulator through a pair of saline-soaked sponge electrodes kept firm by elastic bands.
  For the OW/OB with diagnosis of BE, or food craving, the anode will be placed on the right PFC, F4 position according to the 10-20 international EEG system for electrode placement, while the cathode will be placed on the left PFC, F3 position according to the 10-20 international EEG system for electrode placement.
  Stimulation intensity will be set at 1 milliampere (mA), the duration of stimulation will be 20 min.
  Other Names: Brain Stim
  Arms: BED Active tDCS
Device: BED Sham tDCS — The same electrode placement will be used as in the stimulation conditions (right anodal/left cathodal), but the current will be applied for 30 s and will be ramped down without the participants awareness, and will be held three times a week for six weeks.
  Other Names: Brain Stim
  Arms: BED Sham tDCS

SUMMARY:
The present study grounds on the possible role of hemispheric lateralization in Eating disorders (ED): specifically, hyperactivity of the right frontal regions in Anorexia Nervosa (AN), and hypoactivity of the right frontal regions in Binge Eating Disorder (BED) and food craving behaviors.

Therefore, the investigators hypothesized that active excitatory tDCS over left prefrontal cortex (PFC) (Anode left/cathode right) may aid in altering/resetting inter-hemispheric balance in AN patients, re-establish control over eating behaviors. On the contrary, active excitatory tDCS over right PFC (Anode right/cathode left) may aid in altering/resetting inter-hemispheric balance in BED patients and people with frequent food cravings, decreasing cravings/appetite binge eating behaviors.

DETAILED DESCRIPTION:
The study design is randomized stratified, double blind, add-on, placebo-controlled.

A group of children and adolescents with AN will be selected and randomly assigned to two different conditions: treatment "as usual" plus experimental treatment (active tDCS); treatment "as usual" plus placebo treatment (sham tDCS).

Similarly, a group of children and adolescents with Over-weight/Obesity (OW/OB) and BED will be selected and assigned with randomized stratified sampling to the following conditions: treatment "as usual" plus experimental treatment (active tDCS); treatment "as usual" plus placebo treatment (sham tDCS).

In this project, the investigators will work to understand whether a brain-based treatment, with the use of tDCS, can improve the outcome of patients with eating disorders.

The investigators will test whether tDCS treatment produces improvements in under-eating and over-eating diseases, such us AN and OW/OB with BED and food craving.

Our overarching goal is to provide a scientific foundation for devising new rehabilitation strategies in ED.

ELIGIBILITY:
Inclusion Criteria:

* Under-weight (BMI less than 5th percentile)1 with Clinical diagnosis of AN as described in the 5th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
* Over-weight/Obesity (OW/OB) (BMI above the 85th percentile)1 with diagnosis of BED, or with food craving behaviors
* Ability to give informed consent under parents' surveillance and guidance

Exclusion Criteria:

* Having a comorbidity with an important medical condition;
* Having neurological diseases
* Having Epilepsy o family history of epilepsy
* Pregnant or planning to become pregnant;
* Suicide risk;
* Receiving counseling or psychological therapies during the study;
* Receiving a treatment for an eating disorder in the previous three months before the baseline screening visit.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-07; Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
The primary end-point of the study is the mean change in the Overcontrol composite score of Eating Disorder Inventory - Three (EDI-3) questionnaire, using an approach based on the magnitudes of change. | 6 weeks
  the mean change in the Overcontrol composite score of the EDI-3 questionnaire gives a measure of the basic characteristics of the eating disorders and is a prognostic measure of outcome of eating disorders. Indeed, patterns of treatment response revealed significantly changes in terms of reduced eating disorder symptoms and fewer psychological problems.

SECONDARY OUTCOMES:
The proportion of patients in the two arms with improvement in the total scores of other psychopathological measures as the Yale-Brown-Cornell Eating Disorder Scale (YBC-EDS) questionnaire | 6 weeks
The proportion of patients in the two arms with improvement in the total scores of other psychopathological measures as the BINGE EATING SCALE (BES) questionnaire | 6 weeks
The proportion of patients in the two arms with improvement in the neuropsychological measure of executive control and reward sensitivity by the 'Bechara Iowa Gambling' Task | 6 weeks
The proportion of patients in the two arms with improvement in the neuropsychological measure of the ability to stop by THE STOP-SIGNAL REACTION-TIME (SSRT) task. | 6 weeks
The proportion of patients in the two arms with improvement in the neuropsychological measure of visual attention and task switching by the TRAIL MAKING TEST | 6 weeks
The proportion of patients in the two arms with normalization of different physiological measures specifically the BMI index | 12 months follow up
The proportion of patients in the two arms with normalization of different physiological measures specifically the values of bloody pressure | 12 months follow up
The proportion of patients in the two arms with normalization of different physiological measures specifically the values of cardiac frequency | 12 months follow up
The proportion of patients in the two arms with normalization of different physiological measures specifically the values of body composition | 12 months follow up
In the AN group, significant changes in intra-cortical inhibitory/excitatory motor circuits using paired pulse TMS, measured as SICI/ICF: the ratio between MEPs amplitude (mV) conditioning stimulus and MEPs amplitude test stimulus alone for each ISI. | 6 weeks
In the AN group, significant changes in sensory-motor integration using paired pulse TMS, measured as SICI/ICF: the ratio between MEPs amplitude (mV) conditioning stimulus (electrical stimulation) and MEP amplitude test stimulus alone for each ISI. | 6 weeks
In the AN group, significant changes in cortical oscillatory patterns (synchronization and desynchronization) in theta, alpha and beta frequencies (Hz) over motor and premotor cortex, using TMS-EEG co-registration. | 6 weeks
In the AN group, normalization of endogenous stress response, measured with CAR. | 6 months follow up
In the AN group, significant changes in cortical connectivity, through the analysis of the waveform, latency and cortical distribution of TMS-evoked potentials (TEPs) in micronV, using TMS-EEG co-registration. | 6 weeks
In the AN group, significant changes in cortical reactivity in terms of TMS-evoked potentials (TEPs) amplitude for time domain (micronV) and frequency bands for spatial domain (Hz), using TMS-EEG co-registration. | 6 weeks
In the AN group, significant changes in Cortical Plasticity evoked by repetitive TMS in terms of different MEP amplitude (mV) recorded at different time-points after repetitive TMS perturbations. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Vicari, Study Chair — Bambino Gesù Hospital and Research Institute; Floriana Costanzo, Principal Investigator — Bambino Gesù Hospital and Research Institute
Locations (1):
- Bambino Gesù Hospital and Research Institute, Rome, Italy

REFERENCES:
- [Background] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389
- [Result] Costanzo F, Menghini D, Maritato A, Castiglioni MC, Mereu A, Varuzza C, Zanna V, Vicari S. New Treatment Perspectives in Adolescents With Anorexia Nervosa: The Efficacy of Non-invasive Brain-Directed Treatment. Front Behav Neurosci. 2018 Jul 20;12:133. doi: 10.3389/fnbeh.2018.00133. eCollection 2018. PMID 30083095